CLINICAL TRIAL: NCT03298646
Title: Lidocaine Infusion On Hysteroscopic Media Versus Oral Diclofinac For Pain Relief During Outpatient Hysteroscopy: A Randomized Controlled Trial
Brief Title: Lidocaine Infusion On Hysteroscopic Media Versus Oral Diclofinac For Pain Relief During Outpatient Hysteroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Elsayed Hassan Elbohoty, Assistant professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Hysteroscopy
Record Dates: First submitted 2017-08-30; First posted 2017-10-02 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Nulliparity
MeSH Terms: interventions — Lidocaine; Diclofenac

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lidacaine hydrochloride (Experimental): Adding 10 ml of 2% Lidocaine hydrochloride on hysteroscopic saline media during office hysteroscopy to test its efficacy in reducing pain.
  22 women.
  Interventions: Drug: Lidocaine Hydrochloride
- Diclofenac (Active Comparator): 100 mg Diclofenac oral tablet is administered 1 hour before the procedure to test its efficacy in reducing pain.
  22 women.
  Interventions: Drug: Diclofenac

INTERVENTIONS:
Drug: Lidocaine Hydrochloride — 10 ml of 2% lidocaine on hysteroscopic infusion media during office hysteroscopy.
  Arms: Lidacaine hydrochloride
Drug: Diclofenac — 100 mg Diclofenac oral tablet one hour before the procedure.
  Arms: Diclofenac

SUMMARY:
Lidocaine Infusion On Hysteroscopic Media Versus Oral Diclofinac For Pain Relief During Outpatient Hysteroscopy. A Randomized Controlled Trial.

DETAILED DESCRIPTION:
10 ml of 2% lidocaine hydrochloride added on saline infusion media versus 100 mg diclofenac tablet 1 hour before office hysteroscopy , to test their efficacy in reducing pain .

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-35 years.
* BMI 18.5-30 Kg.
* Nulliparous women assigned for diagnostic hysteroscopy.
* Informed written consent.

Exclusion Criteria:

* Previous cervical surgery.
* Cervical stenosis.
* Known gastritis.
* Recent or active PID.
* Cardiac patients.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Pain reduction using Visual Analogue Scale | 30 minutes
  Efficacy of lidocaine on saline media and oral diclofenac in reducing pain during office hysteroscopy from start of the procedure till 30 minutes after, using visual analogue scale to assess the severity of pain

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams maternity hospital, Cairo, Egypt